CLINICAL TRIAL: NCT06550804
Title: Pilot Trial of a Real-time Electronic Adherence Monitoring Intervention for Antiretroviral Therapy
Brief Title: Testing a Real-time Electronic Antiretroviral Adherence Monitoring Intervention
Acronym: A-TEAM
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023-0873
Record Dates: First submitted 2024-07-05; First posted 2024-08-13 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: HIV Infections; Adherence, Medication
MeSH Terms: conditions — HIV Infections; Medication Adherence

STUDY DESIGN:
Intervention Model Description: One group receives intervention and one groups receives routine care only.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A-TEAM (Experimental): This arm receives the A-TEAM approach where the men, their social support (if they have one), and their case manager participate. If the adherence device identifies non-opening of the device, the men are alerted by text or email the same day. If the device identifies non-opening of the device two days in a row, the social support (or case manager) is notified, and if 7 days of non-opening is detected, the case manager is notified.
  Interventions: Behavioral: A-TEAM
- Control (No Intervention): The men are monitored with the adherence device but there is no intervention on their adherence - they otherwise experience routine care and they don't receive alerts if they the device detects non-openings.

INTERVENTIONS:
Behavioral: A-TEAM — Participants randomized to the intervention arm will receive the proposed intervention, which involves an electronic adherence device called Wisepill and triaged text alerts to the user, the social support, and the case manager for same day, two day, and seven day device non-openings.
  Arms: A-TEAM

SUMMARY:
The investigators propose using an electronic adherence device that is basically a pill container that can alert when it is not opened at a scheduled time. The investigators will use this device to alert the medication user at the time when medication is supposed to be taken if the device did not get opened and a pre-identified social support person or case manager when 2 or 7 consecutive days of nonadherence are detected, respectively. The investigators call our approach "A-Team" (Antiretroviral Therapy Electronic Adherence Monitoring). The aims of this application are to determine the acceptability and feasibility of real-time adherence monitoring in support persons and case managers of African American Men who have sex with Men and to test this approach for these men in a 6-month randomized controlled trial among 54 of these men living with HIV and measure ART adherence and viral suppression (the primary outcome).

DETAILED DESCRIPTION:
African American men who have sex with men (AAMSM) have high HIV infection rates and disproportionate mortality. Critical to ending the HIV epidemic are efforts to reduce HIV transmission by optimizing antiretroviral adherence and suppressing viral load. The investigators propose using responsive electronic adherence monitoring (EAM) in a tiered approach from least to most resource utilization where the EAM device alerts the medication user at the time non-adherence is detected and a pre-identified social support person or case manager when 2 or 7 consecutive days of nonadherence are detected, respectively. The investigators call our approach "A-Team" (Antiretroviral Therapy Electronic Adherence Monitoring) because we provide a team serving a common goal to persons struggling with adherence. This intervention draws on the situated Information Motivation Behavioral Skills Model and is informed by emerging social support literature. Real-time ART adherence monitoring with a triaged response to missed doses informs the patient in real-time of each potential non-adherence event, motivates medication adherence, and positively influences adherence behavioral skills, resulting in viral suppression. This study will be the first to discover how social support persons and case managers perceive this approach, what concerns they may have, and how they respond to one or multiple notifications of missed doses. The aims of this application are to determine the acceptability and feasibility of real-time adherence monitoring in support persons and case managers of AAMSM and to pilot a triaged responsive real-time monitoring adherence intervention for AAMSM. The investigators will implement a 6-month pilot randomized controlled trial among 54 AAMSM living with HIV and measure ART adherence and viral suppression (the primary outcome). Lessons learned from this project may be useful to the field of adherence in these and other persons living with HIV and other diseases.

ELIGIBILITY:
Inclusion Criteria:

Participant inclusion criteria:

* AAMSM >18 years with self-reported HIV infection;
* own a working cell phone;
* on ART for at least 6 months;
* have a case manager willing to participate in the study (for the clinical trial); and
* have suboptimal adherence - either have a detectable viral load in the past 6 months, self-reported <90% adherence based on a 3-item measure or referral by their healthcare provider because of a recognized problem with ART adherence.

For social support persons, participants will:

* report that they have a self-described meaningful relationship with the participant;
* be >18 years of age;
* own a working cell phone and;
* be willing to provide support.

For case managers, participants will have worked with clients with HIV at least 6 months prior to their participation in this study and own a working cell phone.

Exclusion Criteria:

* Not meeting the inclusion criteria
* Not agreeing to informed consent concerning interactions with research team, data collection, and access to medical records.
* Candidates must provide consent to obtain a copy of their viral load results during the 12 months before and following study onset to confirm eligibility and explore long-term follow-up of possible effect.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Viral load suppression | At 6 months after introduction of the intervention.
  We measure HIV viral load

SECONDARY OUTCOMES:
Adherence | At the end of month 1, month 2, month 3, month 4, month 5 and at 6 months
  Real-time and self-reported adherence

CONTACTS AND LOCATIONS:
Overall Officials: Mark Dworkin, MD, Principal Investigator — University of Illinois Chicago
Locations (1):
- University of Illinois Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
As individual participant data might contain identifiers since some data is qualitative, we are undecided on how to share data and will seek guidance if the situation arises.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available for one year after the pilot trial efficacy data are published in a peer-reviewed journal.
Access Criteria: Contact principal investigator with rationale and plan